CLINICAL TRIAL: NCT04801576
Title: In Vivo Assessment of Geno- and Cytotoxicity of Fluoridated Toothpastes and Mouthrinses on Human Buccal Epithelial Cells
Brief Title: In Vivo Assessment of Geno- and Cytotoxicity of Fluoridated Toothpastes and Mouthrinses on Buccal Epithelial Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Principal Investigator, Ema Puizina Mladinić, MD, Principal investigator, University of Split, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EPuizina
Record Dates: First submitted 2021-02-23; First posted 2021-03-17 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: DNA Damage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo mouthrinse (Placebo Comparator): Group that uses just toothpaste without fluoride for 28 days; toothpaste without flouride and mouthrinse without flouride for 28 days; toothpaste with 1050 ppm F and mouthrinse without flouride for 28 days; toothpaste with 1450 ppm F and mouthrinse without flouride for 28 days.
  Interventions: Other: Placebo mouthrinse
- Fluoride in mouthrinses (Experimental): Group that uses just toothpaste without fluoride for 28 days; toothpaste without flouride and mouthrinse with 450 ppm F for 28 days; toothpaste with 1050 ppm F and mouthrinse with 450 ppm F for 28 days; toothpaste with 1450 ppm F and mouthrinse with 450 ppm F for 28 days.
  Interventions: Other: Flouride in mouthrinses

INTERVENTIONS:
Other: Flouride in mouthrinses — Custom made toothpastes and mouthrinses that do or do not contain flouride as sodium fluoride in different concentrations.
  Arms: Fluoride in mouthrinses
Other: Placebo mouthrinse — Mouthrinses without flouride
  Arms: Placebo mouthrinse

SUMMARY:
Buccal cells represent the first barrier to the oral hygiene products' potential toxic effect. The usual concentration of fluoride in toothpastes is 1000/1100 parts per million (ppm F); toothpastes with higher (1500 ppm F) and lower than conventional fluoride levels (around 500 ppm F) are available in many countries. Toothpastes containing higher concentrations of fluoride confer greater protection against caries but at the same time the fluoride is able to induce harmful effects on oral mucosa cells.

The study would include around 40 participants, aged between 20 and 65, divided in two groups. Each group will use fluoride free toothpaste for 28 days, than afterwards group B will get toothpastes (each for 28 days) with no fluoride, 1045 ppm F and 1450 ppm F used together with mouthrinse containing 450 ppm F, while the group A will have everything the same except the mouthrinse that will contain no fluoride - a placebo mouthrinse.

Every 28 days buccal cells samples would be collected from each participant and a Buccal micronucleus cytome assay would be performed according to Nature protocols: Thomas et all.

The aim of this study would be to assess the possible cumulative effect of together use of fluoridated toothpastes and mouthrinses, since population worldwide uses them together without any exact studies about toxicity.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* a sufficient level of education to understand the procedures
* patients not younger than 18 and not older than 65 years
* non-smokers
* patients without exposure to any x-ray examination in last 6 months

Exclusion Criteria:

* subjects with use of any medications
* subjects that use alcohol
* subjects with oral lesions
* subjects with history of chronic health conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related cytotoxic and genotoxic events in buccal cells assessed by buccal cytome micronucleus assay. | 112 days (4 periods of 28 days)
  Method used is Buccal Micronucleus Cytome (BMCyt) assay as minimally invasive method for studying DNA damage, chromosomal instability, cell death and the regenerative potential of human buccal mucosal tissue. This is one of the current established methods for buccal cell collection using a small-headed toothbrush, the generation of a single-cell suspension, slide preparation using cytocentrifugation, fixation and staining using Feulgen and Light Green for both bright field and fluorescence microscopic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Split School of medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tadin A, Gavic L, Govic T, Galic N, Zorica Vladislavic N, Zeljezic D. In vivo evaluation of fluoride and sodium lauryl sulphate in toothpaste on buccal epithelial cells toxicity. Acta Odontol Scand. 2019 Jul;77(5):386-393. doi: 10.1080/00016357.2019.1577988. Epub 2019 Feb 20. PMID 30784350
- [Result] Tadin A, Gavic L, Zeravica A, Ugrin K, Galic N, Zeljezic D. Assessment of cytotoxic and genotoxic effects of conventional and whitening kinds of toothpaste on oral mucosa cells. Acta Odontol Scand. 2018 Jan;76(1):64-70. doi: 10.1080/00016357.2017.1384567. Epub 2017 Sep 29. PMID 28959909
- [Result] Tadin A, Marovic D, Galic N, Kovacic I, Zeljezic D. Composite-induced toxicity in human gingival and pulp fibroblast cells. Acta Odontol Scand. 2014 May;72(4):304-11. doi: 10.3109/00016357.2013.824607. Epub 2013 Aug 22. PMID 23964631
- [Result] Ribeiro DA, Cardoso CM, Yujra VQ, DE Barros Viana M, Aguiar O Jr, Pisani LP, Oshima CTF. Fluoride Induces Apoptosis in Mammalian Cells: In Vitro and In Vivo Studies. Anticancer Res. 2017 Sep;37(9):4767-4777. doi: 10.21873/anticanres.11883. PMID 28870895
- [Result] Thomas P, Holland N, Bolognesi C, Kirsch-Volders M, Bonassi S, Zeiger E, Knasmueller S, Fenech M. Buccal micronucleus cytome assay. Nat Protoc. 2009;4(6):825-37. doi: 10.1038/nprot.2009.53. Epub 2009 May 7. PMID 19444240